CLINICAL TRIAL: NCT06635304
Title: A Retrospective Observational Mono-center Study Of Miniscrews Placement For Orthodontic Anchorage
Brief Title: Miniscrews Placement for Orthodontic Anchorage
Status: Active, not recruiting | Type: Observational
Sponsor: IRCCS San Raffaele (Other)
Responsible Party: Principal Investigator, Simona Tecco, Associate Professor, IRCCS San Raffaele
Other Study IDs: TADs
Record Dates: First submitted 2024-10-06; First posted 2024-10-10 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2024-10

CONDITIONS: Miniscrew Placement; Third Palatal Ruga
Keywords: Miniscrews; Third palatal ruga

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Deep vault: All digital models with deep palatal vault will be included in this group. The depth of the vaults will be assessed according to the Korkhaus index, which sets the cutoff for determining the depth of the palatal vault at 42%. Below this percentage, the vault is considered deep; above this percentage, it is considered flat.
- Flat vault: All digital models with flat palatal vault will be included in this group. The depth of the vaults will be assessed according to the Korkhaus index, which sets the cutoff for determining the depth of the palatal vault at 42%. Below this percentage, the vault is considered deep; above this percentage, it is considered flat.

SUMMARY:
The goal of this retrospective observational mono-center study is to evaluate inter- and intra-operator variability and accuracy in miniscrews placement compared to CBCT-guided planning. The main questions it aims to answer are:

* Is there inter- and intra-operator variability in miniscrews placement?
* Is CBCT-guided placement more accurate than direct technique?
* Is there consistency among operators in identifying the third palatal ruga?
* Is there an influence of palatal vault morphology on these results?

The study will be conducted on a sample of 736 cases, that underwent digital planning for palatal mini-implants with the superimposition between the virtual model of the arch and the CBCT or latero-lateral teleradiography. The sample will be provided by a specialist in the field (Professor Giuseppe Perinetti, Adjunct Professor at Vita-Salute San Raffaele University) in anonymized form. From this sample the virtual models, that meet inclusion and exclusion criteria, will be selected and divided in two subgroups according to the palatal vault morphology (deep/flat) using the Korkhaus Index, which relates the distance between the first molars (specifically between the intersection point of the transverse groove and the buccal groove of each first molar) and the height of the palatal vault (i.e., the length of a vertical line perpendicular to the median palatal suture and the previously drawn line) setting the cutoff to determine the depth of the palatal vault at 42%. Below this percentage, the vault is considered flat; above this percentage, it is considered deep.

The operators involved will be orthodontists with varying levels of experience. At two different times, using Meshmixer software, they will digitally place a miniscrew in the left hemi-palate of each model and identify the most medial and lateral point of third palatal ruga. The placement of the miniscrews will be repeated by the same operators on the same models after a period of time.

Before proceeding with the placement, they will be instructed on the clinical references for positioning palatal mini-implants and on the use of Meshmixer software. Two trial placements will be proposed to make operators familiarize with the software and the described positioning parameters in the presence of an expert clinician.

The most adopted references in the literature, which will be therefore illustrated, are as follows:

* Placement at the third palatal ruga or up to 2 mm posteriorly, specifying that some authors discourage positioning directly over the third palatal ruga due to the risk of incorrect mini-implant angulation during insertion
* A distance from the midline ranging from 3 to 5 mm
* Regarding the inclination of the mini-implant, it was specified that Wilmes and co-authors recommend inserting it perpendicularly to the occlusal plane, although this parameter was not considered; what truly matters is the point where the mini-implant penetrates the bone.

The identification of the third ruga and the positioning of the mini-implant will occur at different times and in random order.

Data collected will be analyzed through statistical methods.

ELIGIBILITY:
Inclusion Criteria:

* Completeness of data and records
* Good quality of available records, particularly models and CBCT
* Healthy patients
* Digital planning performed using CBCT
* Placement of orthodontic mini-implants in the anterior paramedian area of the palate

Exclusion Criteria:

* Craniofacial anomalies and congenital syndromes (such as cleft lip and palate)
* Cysts and tumors of the jaws
* Presence of impacted teeth
* Presence of several palatal ectopias of the teeth

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Data will be collected from patients treated between 2021 and 2024 with an age range of 11 to 55 years with the most represented age group being 12-30 years. The patients underwent only the CBCT-guided digital planning of mini-implant placement performed in compliance with ALADA principle.Therefore, patients may not have subsequently undergone the actual clinical insertion of the miniscrews. The patient data were anonymously collected at Professor Giuseppe Perinetti's private clinic.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2025-01-07 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Inter- and intra-operator variability and accuracy in miniscrews direct placement compared to CBCT-guided planning | Baseline, up to 1 month
  For each model, miniscrew coordinates (as placed by recruited orthodontists) will be recorded. To this purpose, all models will be prepared using Meshmixer software (version 3.5; Autodesk Inc) by positioning the Y-axis reference on the median palatal suture and considering the center of the Cartesian coordinate system at the most distal point of the incisive papilla. Miniscrew position and reference position planned with CBCT will be statistically compared using parametric or non-parametric tests depending on the normality of the data. Miniscrew placement will be repeated on the same models by the same operators within 1 month after.

SECONDARY OUTCOMES:
Consistency among operators in identifying the third palatal ruga | Immediatly after the procedure
  For each model, recruited orthodontists will identify the most medial and the most lateral points of the third palatal ruga.

OTHER OUTCOMES:
Influence of palatal vault morphology on primary and secondary outcome | Through study completion, an average of 6 months
  For each model, palatal vault morphology (deep/flat) will be assessed according to Korkhaus index.

CONTACTS AND LOCATIONS:
Overall Officials: Enrico Gherlone, Study Chair — IRCCS San Raffaele Hospital
Locations (1):
- Dental Clinic, IRCCS San Raffaele Hospital, Milan, Italy, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Hoggan BR, Sadowsky C. The use of palatal rugae for the assessment of anteroposterior tooth movements. Am J Orthod Dentofacial Orthop. 2001 May;119(5):482-8. doi: 10.1067/mod.2001.113001. PMID 11343019
- [Background] Iodice G, Nanda R, Drago S, Repetto L, Tonoli G, Silvestrini-Biavati A, Migliorati M. Accuracy of direct insertion of TADs in the anterior palate with respect to a 3D-assisted digital insertion virtual planning. Orthod Craniofac Res. 2022 May;25(2):192-198. doi: 10.1111/ocr.12525. Epub 2021 Aug 9. PMID 34344059
- [Background] Almeida MA, Phillips C, Kula K, Tulloch C. Stability of the palatal rugae as landmarks for analysis of dental casts. Angle Orthod. 1995;65(1):43-8. doi: 10.1043/0003-3219(1995)0652.0.CO;2. PMID 7726462
- [Background] Cantarella D, Savio G, Grigolato L, Zanata P, Berveglieri C, Lo Giudice A, Isola G, Del Fabbro M, Moon W. A New Methodology for the Digital Planning of Micro-Implant-Supported Maxillary Skeletal Expansion. Med Devices (Auckl). 2020 Mar 18;13:93-106. doi: 10.2147/MDER.S247751. eCollection 2020. PMID 32256130